CLINICAL TRIAL: NCT02736214
Title: Reproductive Life Plan-based Counseling With Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Maja Bodin, PhD-student, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RLP-man-RCT
Record Dates: First submitted 2016-04-01; First posted 2016-04-13 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Sexual Behavior; Lifestyle; Fertility; Pregnancy; Gender Role
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Who Masked: Participant
Masking Description: The randomization was blind to the participants, but they were made aware of their allocation during the intervention

ARMS (2):
- Lifestyle counseling (Experimental): The intervention group answered a baseline questionnaire in the waiting room and received the intervention (Reproductive Life Plan) in addition to standard care.
  Interventions: Behavioral: Reproductive Life Plan (RLP)
- Control group (No Intervention): The control group answered a baseline questionnaire in the waiting room and received standard care.

INTERVENTIONS:
Behavioral: Reproductive Life Plan (RLP) — A structured discussion based on the RLP, including information about reproduction and a brochure with the same information.
  Arms: Lifestyle counseling

SUMMARY:
Many women and men in fertile age are at risk for sexual transmitted infections and unwanted pregnancies, and have insufficient knowledge of health promoting lifestyle prior to conception. There is a need to increase awareness among people in fertile age about how sexual risk-taking and unhealthy lifestyle can negatively affect fertility and pregnancy outcomes. Previous studies on preconception health and care have mainly focused on women. The aim of our study was to investigate if Reproductive Life Plan-based counseling with a midwife could increase men's reproductive knowledge. The second aim was to evaluate men's experiences of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Visitors at drop-in hours at two clinics testing for sexually transmitted infections

Exclusion Criteria:

* Non-Swedish speaking
* Female gender identity

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 229 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2016-04-25 (Actual)

PRIMARY OUTCOMES:
Knowledge of reproduction, measured by a total knowledge score | 2-3 months after the intervention
  Knowledge of reproduction will be measured by knowledge of the following items:
  * the viability of an ovum
  * the viability of sperm
  * how likely it is that a 25-year old women gets pregnant if she has unprotected intercourse at the time of ovulation
  * at what age there is a marked decline in women's ability to become pregnant
  * the proportion of infertility-cases that are caused by a male factor
  * success rate of IVF-treatment
  The outcome will be given as a total score, based on number of correct answers to the items above, and compared to the total score at baseline
Knowledge of lifestyle related factors that can affect fertility, measured by the total number of factors mentioned | 2-3 months after the intervention
  The participants will be asked to mention as many factors as they can remember that
  * can impair male fertility
  * could be modified in the preconception period to increase the chances of conception and having a healthy offspring
  The number of factors mentioned after the intervention will be compared to the number of factors mentioned at baseline

SECONDARY OUTCOMES:
Overall experiences of the intervention (Likert-scale) | 2-3 months after the intervention
  Experience of the intervention is measured on a Likert-scale by the question of
  - The participants overall experience of the intervention (very positive - very negative)
Experience of discussing reproductive life plan (RLP) with a midwife (Likert-scale) | 2-3 months after the intervention
  Experience of discussing RLP with a midwife is measured on a Likert-scale by the question
  - How was the experience of talking to a midwife about the reproductive life plan (very positive - very negative)
Generating new thoughts (Likert-scale) | 2-3 months after the intervention
  If the intervention could generate new thoughts on reproduction is measured on a Likert-scale by the question
  - Has the intervention brought new thoughts about reproduction (In very large extent - in very small extent)
Generating further knowledge seeking (Likert-scale) | 2-3 months after the intervention
  If the intervention could lead to further knowledge seeking is measured on by the question
  - Did the discussion with the midwife lead to a search for more information about reproduction (A lot more - some more - not at all)
Implications for future health care seeking (Likert-scale) | 2-3 months after the intervention
  Whether the availability of discussing RLP with a midwife would be of future interest is measured on a Likert-scale by the question
  - The likelihood of approaching a midwife if more questions about reproduction occured (Very likely - Very unlikely)
Implications for implementing RLP-counseling as a routine (yes/no) | 2-3 months after the intervention
  The acceptance of implementing RLP-counselling as a routine is measured by the question
  - Should midwives or other health care professionals routinely discuss the Reproductive Life Plan with their patients (yes/no)
Likelihood of future lifestyle change (Likert-scale) | 2-3 months after the intervention
  Whether participants would consider making a preconception lifestyle change is measured on a Likert-scale by the question
  - The likelihood among of making a lifestyle change in the future when planning for a pregnancy (Very likely - Very unlikely)
Importance of discussing fertility and preconception health with men (Likert-scale) | 2-3 months after the intervention
  The perceived significance of RLP-counselling is measured on a Likert-scale by the question
  - The importance of informing/educating men about fertility and preconception health issues (Very important - Very unimportant)

CONTACTS AND LOCATIONS:
Overall Officials: Maja Bodin, Principal Investigator — Uppsala University, Sweden; Margareta Larsson, PhD, Study Director — Uppsala University, Sweden
Locations (2):
- Sweden (2):
  - The RFSU clinic, Stockholm
  - Flogsta Mansmottagning, Uppsala

REFERENCES:
- [Background] Warner JN, Frey KA. The well-man visit: addressing a man's health to optimize pregnancy outcomes. J Am Board Fam Med. 2013 Mar-Apr;26(2):196-202. doi: 10.3122/jabfm.2013.02.120143. PMID 23471934
- [Background] Stern J, Larsson M, Kristiansson P, Tyden T. Introducing reproductive life plan-based information in contraceptive counselling: an RCT. Hum Reprod. 2013 Sep;28(9):2450-61. doi: 10.1093/humrep/det279. Epub 2013 Jul 10. PMID 23842564
- [Background] Frey KA, Navarro SM, Kotelchuck M, Lu MC. The clinical content of preconception care: preconception care for men. Am J Obstet Gynecol. 2008 Dec;199(6 Suppl 2):S389-95. doi: 10.1016/j.ajog.2008.10.024. PMID 19081435
- See also: Homepage of Department of Women's and Children's Health, Uppsala University — http://kbh.uu.se